CLINICAL TRIAL: NCT07099352
Title: Efficacy of of Acupuncture Laser Therapy on Neck Pain Severity and Quality of Life in Hemodialysis Patients
Brief Title: Efficacy of of Acupuncture Laser Therapy on Hemodialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, Academic researcher, Sinai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005538
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis
Keywords: Hemodialysis, Acupuncture Laser Therapy

STUDY DESIGN:
Intervention Model Description: This expected prospective randomized control trial study will involve 60 haemodialysis patients with neck pain. The patients in the experimental group (E) will subject, medical treatment besides acupuncture laser therapy. Medical treatment will be used in the control group (C). Pain and quality of life assessment will be used in the assessment of outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efficacy of of Acupuncture Laser Therapy on Hemodialysis (Experimental): This expected prospective randomized control trial study will involve 60 hemodialysis patients with neck pain. The patients in the experimental group (E) will subject, medical treatment besides acupuncture laser therapy. Medical treatment will be used in the control group (C). Pain and quality of life assessment will be used in the assessment of outcome.
  Interventions: Device: Acupuncture Laser Therapy

INTERVENTIONS:
Device: Acupuncture Laser Therapy — Participants will receive low-level laser therapy sessions during dialysis , applied three times per week for 4 weeks to selected treatment areas.

SUMMARY:
This expected prospective randomized control trial study will involve 60 haemodialysis patients with neck pain. The patients in the experimental group (E) will subject, medical treatment besides acupuncture laser therapy. Medical treatment will be used in the control group (C). Pain and quality of life assessment will be used in the assessment of outcome.

DETAILED DESCRIPTION:
The present study will carry out on 60 participants with Haemodialysis that will treat in Hehia hospital that is specialized in physical therapy for Hemodialysis. sixty hemodialysis patients undergoing physical therapy treatments will participate in the study. Their mean age will range from (18-65) years old. The exclusion criteria were as follows: a failure to take part in more than three light therapy sessions; a kidney transplant; and death.

ELIGIBILITY:
Inclusion Criteria:

-Their mean age will range from (18-65) years old.

Exclusion Criteria:

-a failure to take part in more than three light therapy sessions; a kidney transplant; and death.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
change in pain scales | baseline and after 2 weeks of treatment
  visual analogue scale
change in Quality of life scale | baseline and after 2 weeks of treatment
  Chronic neck pain is a common issue among individuals undergoing hemodialysis, often resulting from factors such as poor posture during treatments, muscle tension, and underlying health conditions. Traditional pain management strategies may not always provide adequate relief and can have undesirable side effects, especially in patients with complex medical histories.
change of perceived stress scale | Baseline and after 4 weeks of treatment
  Chronic neck pain is a common issue among individuals undergoing hemodialysis, often resulting from factors such as poor posture during treatments, muscle tension, and underlying health conditions. Traditional pain management strategies may not always provide adequate relief and can have undesirable side effects, especially in patients with complex medical histories.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university- Faculity of physical therapy, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
sixty patients undergoing physical therapy treatments in Hehia hospital will participate in the study. Their mean age will range from (18-65) years old. The exclusion criteria were as follows: a failure to take part in more than three light therapy sessions; a kidney transplant; and death.